CLINICAL TRIAL: NCT07157137
Title: Assessment of the Adherence to a Gluten-free Diet and Nutritional Status of Paediatric Patients With Coeliac Disease
Acronym: CD-PL
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Banaszkiewicz, MD, PhD, Prof., Medical University of Warsaw
Other Study IDs: CD-PL
Record Dates: First submitted 2025-08-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease in Children; Gluten-free Diet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with coealiac disease.: Patients will undergo anthropometric measurements (body weight, height, and thickness of skin folds over the triceps brachii muscle).
  Patient data will be collected during the study, including age, gender, date of coeliac disease diagnosis, duration of gluten-free diet and adherence, history of chronic diseases and congenital defects, medications taken, reported allergies, and family history, with particular emphasis on autoimmune diseases. Guardians/parents of patients under 10 years of age and patients over 10 years of age will be asked to complete a validated Celiac Dietary Adherence Test form. For all patients: IgA tissue transglutaminase antibody levels, aminotransferase activity, complete blood count, and ferritin levels will be measured. An additional 5 ml of venous blood will be collected to measure albumin, folic acid, vitamins B12, A, E, 25-OH vitamin D, and a lipid profile. Additionally, a urine and stool sample will be collected to measure gluten immunogenic peptides.

SUMMARY:
Although a gluten-free diet (GFD) is essential for patients with coeliac disease (CD), many do not follow it strictly. Exposure to gluten causes villous atrophy, can deteriorate nutritional status, and can lead to deficiencies. The ESPGHAN recommends combining multiple methods to assess GFD adherence. The Celiac Dietary Adherence Test (CDAT) and measuring the gluten immunogenic peptide in urine (uGIP) or stool (sGIP) were suggested.

This study aims to evaluate and compare the usefulness of an adapted CDAT, the rapid tests for detecting uGIP and sGIP, for assessing adherence to a GFD in children with CD. Additionally, we will assess these children's nutritional status.

Patients, aged 2-18 years, diagnosed with CD, who have been on a GFD for at least 6 months, will be included. Clinical characteristics and anthropometric measurements will be recorded. The adapted CDAT form will be applied. A single urine and stool samples will be collected immediately, and rapid tests for the detection of GIP will be performed. The serum levels of anti-transglutaminase antibodies (IgA), albumin, ferritin, folate, vitamins B12, A, E, 25-OH vitamin D, blood count and lipid profile will be measured.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of coeliac disease according to the European Society of Pediatric Gastroenterology and Nutrition (ESPGHAN) criteria,
* age from 2 to 18 years of age,
* gluten-free diet use for at least 6 months,
* consent from legal guardians (and the child in case of patients ≥16 years of age) to participate in the study.

Exclusion criteria:

* under 2 years of age and over 18 years of age,
* immunoglobulin A deficiency,
* inflammatory bowel diseases,
* gastrointestinal bleeding or other active bleeding,
* gastric and/or duodenal ulcers,
* liver failure,
* heart failure according to the NYHA II-IV scale,
* acute and chronic renal failure,
* cancer,
* after hematopoietic stem cell transplantation,
* whose legal guardians did not consent to participate in the study,
* who did not consent to participate in the study (applies to patients ≥ 16 years of age).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Polish children with CD.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to a gluten-free diet - the Celiac Dietary Adherence Test. | January 2026 - June 2027
  Adherence to the gluten-free diet will be assessed based on positive results in the Celiac Dietary Adherence Test questionnaire.
Adherence to the gluten-free diet - the gluten immunogenic peptide in urine. | January 2026 - June 2027
  Adherence to the gluten-free diet will be assessed based on positive results in the gluten immunogenic peptide in urine (uGIP).
Adherence to the gluten-free diet - the gluten immunogenic peptide in stool. | January 2026 - June 2027
  Adherence to the gluten-free diet will be assessed based on positive results in the gluten immunogenic peptide in stool (sGIP).
Comparison of methods | January 2026 - June 2027
  The results of CDAT questionnaire, uGIP and sGIP will be compared to the standard IgA tissue transglutaminase antibody test. Intra-assay agreement will be assessed using the McNemary test. Measures of test quality (sensitivity, specificity, positive and negative predictive values) will be calculated.

SECONDARY OUTCOMES:
The nutritional status of Polish children with coeliac disease | January 2026 - June 2027
  The nutritional status of Polish children with coeliac disease will be assessed by analysing the anthropometric measurements and laboratory tests performed. The results obtained will be compared with data obtained for the general population.